CLINICAL TRIAL: NCT06092710
Title: Predictive Value of OSA Based on the Evaluation of the Subjective Feeling of the Air Flow Through Airways, a Randomized Controlled Study
Brief Title: Predictability of OSA With a Subjective Screening Scale (OSASSS1)
Acronym: OSASSS1
Status: Completed | Type: Observational
Sponsor: Center for Sleep Medicine - Clinique André Renard (Other)
Collaborators: PIRON Alain, Osteopath - physiotherapist (Unknown); LACROIX Alain, neurologist, MD, PhD (Unknown); CHAKAR Bassam, neurologist, MD, PhD (Unknown)
Responsible Party: Principal Investigator, GARCION Cédric, Principal Investigator, Center for Sleep Medicine - Clinique André Renard
Other Study IDs: OSASSS1
Record Dates: First submitted 2023-10-07; First posted 2023-10-23 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea; OSA
Keywords: obstructive sleep apnea; OSA; obstructive sleep apnea syndrome; sleep disorder; upper airways resistance syndrome UARS; subjective scale of air flow
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group with PSG and sleep survey: the study group will be recruited after their polysomnography but before its results, so patients and investigators will not have any data about Apnea Hypopnea Index (AHI) and sleep survey. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  Interventions: Diagnostic Test: neuro-sensorial subjective evaluation of the airways collapsibility
- control group with sleep survey: the control group will be recruited after a sleep survey with no sleep disorder. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  Interventions: Diagnostic Test: neuro-sensorial subjective evaluation of the airways collapsibility

INTERVENTIONS:
Diagnostic Test: neuro-sensorial subjective evaluation of the airways collapsibility — verbal and manual guidance of subjects from a therapist to experiment the subjective perception of the air flow through their airways and airways collapsibility
  Other Names: subjective perception scale of the air flow through airways; subjective perception of the air flow protocol; protocol of subjective perception of airways collapsibility; subjective perception scale of airways collapsibility

SUMMARY:
the study aims to evaluate the accuracy correlation between subjective perception of the air flow through airways from patients and survey and/or polysomnography they spent, using a brief clinical protocol they answered with a manual therapist

DETAILED DESCRIPTION:
The subjects in the study are 18 to 77 years old and present the following conditions:

* polysomnography and sleep survey realized at the Center for Sleep Medicine André RENARD, without any informations of the results for the experience group
* sleep survey with no sleep trouble found for the control group

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18 to 77 years old
* subjects who have performed a PSG at the sleep medicine center André Renard for the study group
* subjects with no sleep disorder on sleep survey for the control group
* Subjects who agree to comply with the requirements of the study.
* Subjects who are of age (and know how to read and write) who have given their informed, explicit consent in advance to any procedure related to the trial, the study or the investigation conducted on human beings, with the objective of developing knowledge specific to the exercise of health care professions, as set out in Royal Decree No. 78 of 10 November 1967 on the practice of the health care professions (Act of 27 December 2005)

Exclusion Criteria:

* subjects with acute infections
* subjects with trauma within the last 72 hours
* subjects who already benefit from OSA treatment
* subjects with known perceptual disorders, for example post-stroke
* subjects with current or recent chemotherapy and radiotherapy treatment
* Pregnant women
* Criteria related to prior or concurrent treatments:

Treatment with antipsychotics, anxiolytics, soporifics or muscle relaxants started within the two months preceding the study.

Treatment with intraoral implants during the study or in the two months preceding the study

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with OSA objectified after polysomnography, sleepiness Epworth scale, fatigue Pichot scale, and subjects without OSA specified by negativation at sleepiness Epworth scale, fatigue Pichot scale, Berlin questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain LACROIX, Neurologist, PhD, Study Chair — Center of Sleep Medecine - Clinique André Renard
Locations (1):
- Centre de médecine du sommeil- Clinique André Renard, Herstal, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared after anonymization of the subjects
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: November 2023 to December 2024
Access Criteria: Any approved researcher or reviewer who needs the data to compare, experiment or monitor the study for an official agency or international publication will be able to contact us and obtain the study data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place by invitation to the sleep laboratory of the Clinique Andre Renard, from 01/01/2023 to 31/12/2023 for the study and control groups.
  study group determined by 3 neurologists after analysis of their polysomnography to form subgroups with mild, moderate and severe OSA. control group determined by questionnaires sent to subjects. The questionnaires had to have responses below the scores for suspected sleepiness or fatigue in order to be included in the control group.
Period: Overall Study
Arm/Group | Study Group With PSG and Sleep Survey | Control Group With Sleep Survey
Started | 52 | 60
Completed | 52 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 52 participants in the study group with PSG and sleep survey: 11 with a negative diagnosis for sleep apnea 9 with a positive diagnosis of mild OSA 18 with a positive diagnosis of moderate OSA 14 with a positive diagnosis of severe OSA 60 participants in the control group with sleep survey: all negative for suspicion of sleep apnea with 4 questionnaires these are not results or a conclusion drawn from the results, but a factual description of the composition of the groups as requested.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group With PSG and Sleep Survey | Control Group With Sleep Survey | Total
Number analyzed (Participants) | 52 | 60 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 57 | 104
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.8) | 41.8 (12.8) | 44.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 40 | 65
  Male | 27 | 20 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 52 | 60 | 112
Body Mass Index Body Mass Index (BMI) units: kg/m2 Mean (Standard Deviation) [Mean (Standard Deviation); unit: kg/m2] | 29.3 (5.8) | 22.8 (3.3) | 25.8 (5.7)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0 (no chance of dozing) to 3 (high chance of dozing). When you finish the test, add up the values of your responses. Your total score is based on a scale of 0 to 24.
  * Below 8: you have no sleep debt.
  * From 9 to 14: you have a sleep debt; review your habits.
  * over 15: you are showing signs of excessive daytime sleepiness, medical attention is required
  units on a scale | 10.8 (5.35) | 5.6 (2.2) | 8 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Test of Perception of Variations in the Passage of an Airflow Through the Rhino-oro-pharyngeal Passages According to the Categories of Items Used in the OSASSS Subjective Perception Scale
Description: In this study, we set out to create a scale of subjective perception of airflow. Assessment of subjects' perception of airflow using different positions or maneuvers: responses are scored for perceived ease of airflow.
  Items will be assigned "0" if they feel no expected change in airflow due to the maneuver up to "+1" if they feel a variation corresponding to the maneuver. Summed together, they define a score by item category (ST):
  * "constraining" (ST1: min= 0/Max= 4: dorsal decubitus "0/1", modified state of consciousness "0/1", cephalic flexion "0/1", tongue high to low position "0/1")
  * "facilitating" (ST2: min= 0/max=3: mandibular advancement "0/1", cephalic extension "0/1", nasal dilatation "0/1") to then assess whether the sensation of "facilitated or constrained" variation in the passage of air (ST1+ST2: min=0/max=7) is statistically significant for each group of participants compared to the absence of sensation of variation.
Time Frame: during the clinical protocol, about 15 to 20 minutes
Population: Discrete grouping variables :
  healthy patients (= non CHR control patients and normal CHR patients)
  - STATUS 3: 2 categories: non-OSA (control patients and non-OSA CHR patients) and OSA patients (= CHR patients affected to varying degrees)
Measure: Median (99% Confidence Interval); unit: score on a scale
Arm/Group | Study Group With PSG and Sleep Survey | Control Group With Sleep Survey
Number analyzed (Participants) | 52 | 60
score on a scale | 5 [2 to 6] | 4 [0 to 7]
Statistical Analysis 1: Comparison: Study Group With PSG and Sleep Survey vs Control Group With Sleep Survey; Non-parametric tests on patient sensitivity, given the non-normal distribution, (based on the median of the data) were applied to analyse the diﬀerences between the groups (ST1+ ST2 according to the STATUS3 and STATUS4 classification criteria). To analyse any diﬀerences in sensitivity between patient groups, Kruskal-Wallis tests were applied. In this type of analysis, having a p-value greater than 1% and ideally greater than 5% would indicate the absence of diﬀerences between groups; Test type: Other — Then, to see if the median of a particular group is diﬀerent from 0 (= no sensitivity: not feeling the diﬀerences in airflow induced by the diﬀerent tests given by the operator), Wilcoxon tests were performed on each group of data. If the p-value is small (less than 5%, ideally less than 1%), the null hypothesis that the score is identical to 0 is rejected; p = 0.05572, Kruskal-Wallis
Statistical Analysis 2: Comparison: Study Group With PSG and Sleep Survey; to see if the median of a particular group is diﬀerent from 0 (= no sensitivity: not feeling the diﬀerences in airflow induced by the diﬀerent tests given by the operator), Wilcoxon tests were performed on each group of data. If the p-value is small (less than 5%, ideally less than 1%), the null hypothesis that the score is identical to 0 is rejected. In this case, it means that the patients in the test group feel the diﬀerences in airflow depending on their position; Test type: Other — Wilcoxon tests were performed on each group of data. If the p-value is small (less than 5%, ideally less than 1%), the null hypothesis that the score is identical to 0 is rejected; p < 0.0000008, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group With Sleep Survey; [analysis description as in outcome 1, analysis 2]; Test type: Other — Wilcoxon tests were performed on each group of data. If the p-value is small (less than 5%, ideally less than 1%), the null hypothesis that the score is identical to 0 is rejected. In this case, it means that the patients in the test group feel the diﬀerences in airflow depending on their position; p < 0.0000001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Predictability of OSA Based on a Score Using Subjective Perception of Airway Collapsibility Between OSA and Control Subjects to Validate a Clinical Screening Tool
Description: In this study, we set out to create a scale, so we can only describe what we did.
  score by item category (ST):
  * ST1+ST2 (min=0/max=10) corresponds to the sensitivity of "facilitated or constrained" variation in the passage of air.
  * ST3: (min=0/max=3) corresponds to the practitioner's palpation of a synchronous contraction of the floor of the mouth (ventilatory defense sign) and sound turbulence on inspiration
  * ST4 (min=0/max=2) corresponds to lingual posture in supine position (aggravating if low)
  * ST5 (min=0/max=5) corresponds to patients' subjective perception of easy nasal ventilation, snoring, daytime ventilatory mode and nocturnal ventilatory mode
  * ST6 (min=0/max=3) corresponds to the teeth-skeletal class, tonsil grades and Mallampati stages
  * Epworth (min=0/max=2) corresponds to suspected sleep debt
  * FFF (min=0/max=1) corresponds to suspected fatigue SFI (min=0/max=13) corresponds to ST1+ST2+ST3 SFT (min=0/max=26) corresponds to SFI+ST4+ST5+ST6+Epworth+FFF
Time Frame: during the examination and the OSASSS protocol (15 to 20 min)
Population: free-OSA subjects from the CHR (n=11) were excluded from the study group because they had sleep disorders other than OSA
Measure: Mean (99% Confidence Interval); unit: score on a scale
Arm/Group | Study Group With PSG and Sleep Survey | Control Group With Sleep Survey
Number analyzed (Participants) | 41 | 60
score on a scale | 8.63 [7.84 to 9.43] | 5.92 [5.27 to 6.58]
Statistical Analysis 1: Comparison: Study Group With PSG and Sleep Survey vs Control Group With Sleep Survey; Parametric tests on the prediction of patients' pathological status with SFI (Intermediate Final Score) For these analyses, as the SFI score follow a normal distribution, ANOVAs (analyses of variance) were performed. For discrete variables with more than 2 levels of value, a post-hoc 2-to-2 comparison analysis was performed (Tukey) to see which level of the variable diﬀered from one another; Test type: Superiority; p = 0.00000106, ANOVA — Confidence level used: 0.95 Tukey multiple comparisons of means (95% family-wise confidence level)
Statistical Analysis 2: Comparison: Study Group With PSG and Sleep Survey vs Control Group With Sleep Survey; Parametric tests on the prediction of patients' pathological status with SFT score (Final Total score): For these analyses, as SFT score follow a normal distribution, ANOVAs (analyses of variance) were performed. For discrete variables with more than 2 levels of value, a post-hoc 2-to-2 comparison analysis was performed (Tukey) to see which level of the variable diﬀered from one another; Test type: Superiority; p = 0000000048, ANOVA — Confidence level used: 0.95 Tukey multiple comparisons of means (95% family-wise confidence level)
Statistical Analysis 3: Comparison: Study Group With PSG and Sleep Survey vs Control Group With Sleep Survey; Determination of cut-oﬀ values for SFI: The Cutoﬀ_final txt file includes the various sensitivity and specificity calculations as well as the Youden index in order to determine the best cut-oﬀ value (largest Youden). The ROC curves allow the values in the file to be appreciated graphically; Test type: Superiority; p = 0.00000077, Fisher Exact; Odds Ratio (OR) = 8.73
Statistical Analysis 4: Comparison: Study Group With PSG and Sleep Survey vs Control Group With Sleep Survey; Determination of cut-oﬀ values for SFT: The Cutoﬀ_final txt file includes the various sensitivity and specificity calculations as well as the Youden index in order to determine the best cut-oﬀ value (largest Youden). The ROC curves allow the values in the file to be appreciated graphically; Test type: Superiority; p = 0.00000069, Fisher Exact; Odds Ratio (OR) = 9.37

3. Secondary Outcome: Predictive Value on the Severity of OSA of the Subjective Upper Airway Collapsibility Perception Scale
Description: Objective: to determine an intermediate final score (IFS) and total final score (TFS) threshold for classifying the severity of OSA in at-risk subjects. The questionnaire comprises 18 questions relating to upper airway collapsibility. Each item concerns the aggravating or facilitating factors perceived by the patient or therapist during the clinical maneuvers used to obtain the IFS. To obtain the TFS, we add items concerning factors known to be unfavorable to upper airway patency (snoring, mouth ventilation, tonsils, dento-skeletal class, etc.), as well as two questionnaires used in the sleep laboratory at the André Renard Clinic (Epworth sleepiness scale and FFF questionnaire). IFS: min=0/max=13. TFS: min= 0/max=26. The higher the score, the greater the risk of OSA. Clinically, the scale is designed to perform the IFS, giving a score out of 13. Then, if the score is above the first cut-off point, the questionnaire is completed to establish the TFS out of 26.
Time Frame: during the examination protocol, about 15 to 20 minutes
Population: 4 categories:
  * control patients,
  * mild symptom patients (CHR SL),
  * moderate symptom patients (CHR SM)
  * severe symptom patients (CHR SS) free-OSA patients from the CHR study group (n=11) were excluded because they had sleep pathologies other than OSA
  Parametric tests on the prediction of patients' pathological status (SFI and SFT scores):
  ANOVAs were performed. For discrete variables with more than 2 levels of value , a post-hoc 2-to-2 comparison analysis was performed (Tukey).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Control Group: the control group will be recruited after a sleep survey with no sleep disorder. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  neuro-sensorial subjective evaluation of the airways collapsibility: verbal and manual guidance of subjects from a therapist to experiment the subjective perception of the air flow through their airways and airways collapsibility Overall Number of Participants Analyzed: 60
- Mild Symptom Patients (=CHR SL): the study group will be recruited after their polysomnography but before its results, so patients and investigators will not have any data about Apnea Hypopnea Index (AHI) and sleep survey. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  neuro-sensorial subjective evaluation of the airways collapsibility: verbal and manual guidance of subjects from a therapist to experiment the subjective perception of the air flow through their airways and airways collapsibility Overall Number of Participants Analyzed: 9
- Moderate Symptom Patients (= CHR SM): the study group will be recruited after their polysomnography but before its results, so patients and investigators will not have any data about Apnea Hypopnea Index (AHI) and sleep survey. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  neuro-sensorial subjective evaluation of the airways collapsibility: verbal and manual guidance of subjects from a therapist to experiment the subjective perception of the air flow through their airways and airways collapsibility Overall Number of Participants Analyzed: 18
- Severe Symptom Patients (=CHR SS): the study group will be recruited after their polysomnography but before its results, so patients and investigators will not have any data about Apnea Hypopnea Index (AHI) and sleep survey. they will experiment their subjective perception of air flow through their airways with the guidance of a manual therapist during a 15 minutes protocol
  neuro-sensorial subjective evaluation of the airways collapsibility: verbal and manual guidance of subjects from a therapist to experiment the subjective perception of the air flow through their airways and airways collapsibility Overall Number of Participants Analyzed: 14
Arm/Group | Control Group | Mild Symptom Patients (=CHR SL) | Moderate Symptom Patients (= CHR SM) | Severe Symptom Patients (=CHR SS)
Number analyzed (Participants) | 60 | 9 | 18 | 14
score on a scale
  intermediate final score (IFS) | 5.92 [5.26 to 6.59] | 8.78 [7.06 to 10.49] | 8.47 [7.26 to 9.69] | 8.75 [7.37 to 10.13]
  total final score (TFS) | 8.26 [7.34 to 9.18] | 12.89 [10.52 to 15.26] | 12.33 [10.66 to 14.01] | 13.61 [11.71 to 15.51]
Statistical Analysis 1: Comparison: Control Group vs Mild Symptom Patients (=CHR SL); Parametric tests on the prediction of patients' pathological status (SFI and SFT scores): For these analyses, as the SFI and SFT scores follow a normal distribution, ANOVAs (analyses of variance) were performed. For discrete variables with more than 2 levels of value (STATUS4), a post-hoc 2-to-2 comparison analysis was performed (Tukey) to see which level of the variable diﬀered from one another; Test type: Superiority; p = 0.0142266, TUKEY TEST
Statistical Analysis 2: Comparison: Control Group vs Moderate Symptom Patients (= CHR SM); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0023308, TUKEY TEST
Statistical Analysis 3: Comparison: Control Group vs Severe Symptom Patients (=CHR SS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0023308, TUKEY TEST
Statistical Analysis 4: Comparison: Mild Symptom Patients (=CHR SL) vs Moderate Symptom Patients (= CHR SM); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9915779, TUKEY TEST
Statistical Analysis 5: Comparison: Mild Symptom Patients (=CHR SL) vs Severe Symptom Patients (=CHR SS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9999943, TUKEY TEST
Statistical Analysis 6: Comparison: Moderate Symptom Patients (= CHR SM) vs Severe Symptom Patients (=CHR SS); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9905111, TUKEY TEST

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Study Group With PSG and Sleep Survey | Control Group With Sleep Survey
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/60
Other Adverse Events (participants affected / at risk) | 0/52 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT06092710/Prot_SAP_ICF_002.pdf